CLINICAL TRIAL: NCT07007793
Title: A Randomised, Double-Blind, Placebo-Controlled, Parallel-Group Study to Assess the Efficacy and Safety of Baxdrostat in Adult Participants With Primary Aldosteronism
Brief Title: A Study to Assess Efficacy and Safety of Baxdrostat in Participants With Primary Aldosteronism
Acronym: BaxPA
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: D6974C00001
Record Dates: First submitted 2025-05-16; First posted 2025-06-06 (Actual); Last update posted 2026-01-14 (Actual); Status verified 2025-12

CONDITIONS: Primary Hyperaldosteronism
Keywords: Primary hyperaldosteronism; Primary aldosteronism; PA; Baxdrostat; CIN-107; Aldosterone
MeSH Terms: conditions — Hyperaldosteronism

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Baxdrostat (Experimental): Baxdrostat administered orally, once daily (QD).
  Interventions: Drug: Baxdrostat
- Placebo (Placebo Comparator): Matching placebo administered orally, once daily (QD).
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Baxdrostat — Baxdrostat tablet administered orally, once daily (QD).
  Other Names: CIN-107
  Arms: Baxdrostat
Drug: Placebo — Placebo tablet matching baxdrostat, administered orally, once daily (QD).
  Arms: Placebo

SUMMARY:
This is a Phase III, multicentre, randomised, double-blind, placebo-controlled, parallel-group study to evaluate the safety, tolerability, and efficacy of baxdrostat versus placebo, on the reduction of Seated Blood Pressure (SBP) and achieving normalization of the Renin Angiotensin Aldosterone System (RAAS) in approximately 180 participants ≥ 18 years of age with Primary Aldosteronism (PA), with or without prior treatment with Mineralocorticoid Receptor Antagonists (MRAs) or potassium-sparing diuretics.

Baxdrostat (or placebo) will be administered once daily, up-titrated after 2 weeks based on clinical response and tolerability.

The study is planned to be conducted globally in approximately 90 study centres and 12 countries.

ELIGIBILITY:
Inclusion Criteria:

* Male or female participants must be ≥ 18 years of age
* Participants with a documented diagnosis of PA that fulfils the criteria defined in the 2016 or 2025 Endocrine Society Guidelines.
* Participants willing and able to cease dosing of MRA or potassium sparing diuretics per study requirement for participants taking an MRA or potassium sparing diuretic at Screening.
* eGFR ≥ 45 mL/min/1.73m2 at Screening
* Serum potassium level ≥ 3.0 and < 5.0 mmol/L at Screening determined as per the central laboratory.
* Have a stable regimen of antihypertensive medications for at least 4 weeks prior to randomisation
* Mean seated SBP on AOBPM of ≥ 135 mmHg and ≤ 170 mmHg and mean DBP of

  ≤ 105 mmHg.
* Serum potassium (local lab) > 3.0 mmol/L at randomization.

Exclusion Criteria:

- If not taking an MRA or potassium sparing diuretic at Screening: Mean seated SBP > 170 mmHg or mean seated DBP >105 mmHg (on AOBPM).

If taking an MRA or potassium sparing diuretic at Screening: Mean seated SBP > 160 mmHg or mean seated DBP ≥ 100 mmHg.

* Previous surgical intervention for an adrenal adenoma or have a planned adrenalectomy, renal nerve denervation, or adrenal ablative procedure during the course of the study.
* Has the following known secondary causes of HTN: renal artery stenosis, uncontrolled or untreated hyperthyroidism, uncontrolled or untreated hypothyroidism, pheochromocytoma, Cushing's syndrome, aortic coarctation.
* Serum sodium level < 135 mmol/L at Screening, determined as per central laboratory.
* New York Heart Association functional HF class IV at Screening.
* Persistent atrial fibrillation.
* Treatment with any MRA or potassium-sparing diuretic within 2 weeks prior to Randomisation.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 180 (Estimated)
Dates: Start 2025-08-07 (Actual); Primary Completion 2028-02-18 (Estimated); Study Completion 2028-02-18 (Estimated)

PRIMARY OUTCOMES:
Change from baseline in seated Systolic Blood Pressure (SBP) at Week 8 | At week 8
  To assess the effect of baxdrostat versus placebo on seated Systolic Blood Pressure (SBP) at Week 8
Achieving normalization of the Renin Angiotensin Aldosterone system (RAAS) at week 8 | At week 8
  To assess the effect of baxdrostat versus placebo on achieving normalization of the Renin Angiotensin Aldosterone system (RAAS) at week 8, in participants with dysregulated RAAS at baseline

SECONDARY OUTCOMES:
Change from Randomised withdrawal (RWD) baseline (Week 44) in seated Systolic Blood Pressure (SBP) at Week 52 | At week 52
  To assess the effect of baxdrostat versus placebo on seated Systolic Blood Pressure (SBP) 8 weeks after Randomised withdrawal (RWD)
Percent change from RWD baseline (Week 44) in Plasma Renin Activity (PRA) at Week 52 | At week 52
  To assess the effect of baxdrostat versus placebo on the percent change in PRA 8 weeks after RWD
Achieving serum potassium ≥ 3.7 mmol/L without potassium supplementation at Week 8 in participants with serum potassium < 3.7 mmol/L or potassium supplementation at baseline | At week 8
  To assess the effect of baxdrostat versus placebo on achieving serum potassium ≥ 3.7 mmol/L without potassium supplementation at Week 8 in participants with serum potassium < 3.7 mmol/L or potassium supplementation at baseline
Percent change from baseline in PRA at Week 8 | At week 8
  To assess the effect of baxdrostat versus placebo on the percent change from baseline in PRA at Week 8
Achieving 24-hour urine aldosterone < 10 μg at Week 8 in participants with 24-hour urine aldosterone ≥ 10 μg at baseline | At week 8
  To assess the effect of baxdrostat versus placebo on achieving 24-hour urine aldosterone < 10 μg at Week 8 in participants with 24-hour urine aldosterone
  ≥ 10 μg at baseline
Percent change from baseline in 24-hour urine albumin at Week 8 | At week 8
  To assess the effect of baxdrostat versus placebo on 24-hour urine albumin at Week 8

OTHER OUTCOMES:
Number of participants with adverse events (AEs) | up to 54 weeks
  To assess the safety and tolerability of baxdrostat. Occurrence of Adverse Events (AEs), Serious Adverse Events (SAEs), deaths, AEs leading to discontinuation of IMP and adverse events of special interest (AESIs) (hyperkalemia and hyponatremia)

CONTACTS AND LOCATIONS:
Locations (77):
- United States (19):
  - Research Site, Los Angeles, California
  - Research Site, San Francisco, California
  - Research Site, Farmington, Connecticut
  - Research Site, Chicago, Illinois
  - Research Site, Springfield, Illinois
  - Research Site, Baltimore, Maryland
  - Research Site, Boston, Massachusetts
  - Research Site, Ann Arbor, Michigan
  - Research Site, Rochester, Minnesota
  - Research Site, Olive Branch, Mississippi
  - Research Site, Kansas City, Missouri
  - Research Site, New York, New York
  - Research Site, Cleveland, Ohio
  - Research Site, Columbus, Ohio
  - Research Site, Bethlehem, Pennsylvania
  - Research Site, Philadelphia, Pennsylvania
  - Research Site, Columbia, South Carolina
  - Research Site, Brownsville, Texas
  - Research Site, Dallas, Texas
- Australia (3):
  - Research Site, Brisbane
  - Research Site, Clayton
  - Research Site, Perth
- Canada (4):
  - Research Site, Calgary, Alberta
  - Research Site, Ottawa, Ontario
  - Research Site, Toronto, Ontario
  - Research Site, Montreal, Quebec
- China (9):
  - Research Site, Beijing
  - Research Site, Changsha
  - Research Site, Chengdu
  - Research Site, Chongqing
  - Research Site, Nanjing
  - Research Site, Shanghai
  - Research Site, Tianjin
  - Research Site, Wuhan
  - Research Site, Xianyang
- France (6):
  - Research Site, Amiens
  - Research Site, Bois-Guillaume
  - Research Site, Bordeaux
  - Research Site, Lille
  - Research Site, Marseille
  - Research Site, Paris
- Germany (6):
  - Research Site, Berlin
  - Research Site, Düsseldorf
  - Research Site, Kaiserslautern
  - Research Site, München
  - Research Site, Reinfeld (Holstein)
  - Research Site, Würzburg
- India (5):
  - Research Site, Belagavi
  - Research Site, Delhi
  - Research Site, Hyderabad
  - Research Site, Kolkata
  - Research Site, Mumbai
- Italy (5):
  - Research Site, Bologna
  - Research Site, Brescia
  - Research Site, Florence
  - Research Site, Milan
  - Research Site, Torino
- Japan (7):
  - Research Site, Kawasaki-shi
  - Research Site, Kodaira-shi
  - Research Site, Minatoku
  - Research Site, Ōta-ku
  - Research Site, Shinjuku-ku
  - Research Site, Yokohama
  - Research Site, Yufu-shi
- Spain (3):
  - Research Site, Barcelona
  - Research Site, Madrid
  - Research Site, Seville
- Taiwan (6):
  - Research Site, Kaohsiung City
  - Research Site, Taichung
  - Research Site, Taipei
  - Research Site, Taoyuan District
  - Research Site, Yunlin
  - Research Site, Zhubei
- United Kingdom (4):
  - Research Site, Cambridge
  - Research Site, Cardiff
  - Research Site, Dundee
  - Research Site, London

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers can request access to anonymized individual patient-level data from AstraZeneca group of companies sponsored clinical trials via the request portal Vivli.org. All requests will be evaluated as per the AZ disclosure commitment:
  https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
  "Yes", indicates that AZ are accepting requests for IPD, but this does not mean all requests will be approved.
Supporting Information: Study Protocol, SAP
Time Frame: AstraZeneca will meet or exceed data availability as per the commitments made to the EFPIA/PhRMA Data-Sharing Principles. For details of our timelines, please refer to our disclosure commitment at:
  https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
Access Criteria: When a request has been approved AstraZeneca will provide access to the anonymized individual patient-level data via secure research environment Vivli.org. A Signed Data Usage Agreement (non-negotiable contract for data accessors) must be in place before accessing requested information.
URL: https://vivili.org/